CLINICAL TRIAL: NCT03160443
Title: Impact of Neuropsychological Alteration of Decision-making Abilities on the Functioning of Patients With Eating Disorders
Acronym: NEUROPSY_TCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: INSERM 1061, " Neuropsychiatry: epidemiological and clinical research", Montpellier (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9804
Record Dates: First submitted 2017-05-11; First posted 2017-05-19 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Eating Disorder
Keywords: Anorexia nervosa; Bulimia; Binge eating disorders; Neuropsychology; Neurocognition; Daily functioning
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia; Binge-Eating Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Other): All participants performed the same evaluation: clinical and neuropsychological assessment.
  All of them are patients with an eating disorder.
  Interventions: Behavioral: Ambulatory cares in a day-hospital (University Hospital of Montpellier) specialized in the evaluation of eating disorders

INTERVENTIONS:
Behavioral: Ambulatory cares in a day-hospital (University Hospital of Montpellier) specialized in the evaluation of eating disorders — All patients assessed in the day-hospital will performed the same evaluation :
  * Blood sampling
  * Calorimetry
  * Osteodensitometry
  * Psychiatric assessment
  * Endocrinologic assessment
  * Dietetic assessment
  * Neuropsychological assessment
  * Self-questionnaires
  With the patient agreement, a biological collection will be constituted. The objective is the subsequent study of biological factors involved in eating disorders (in particular genetic factors)

SUMMARY:
Eating disorders are multifactorial disorders currently conceptualized in a biopsychosocial model, but pathophysiology remains relatively unknown, and robust etiological models to guide treatment are therefore lacking. Different endophenotypes and neurocognitive vulnerability factors have been found in eating disorders including decision making abnormalities. The investigators hypothesize that decision making abnormalities are associated with a lower level of functioning and quality of life which could lead to social and interpersonal difficulties. The investigators also hypothesize that these anomalies are associated with a particular clinical profile (more restrictive profile, more hyperactivity, less insight on the disease and desire for care ...).

DETAILED DESCRIPTION:
The investigators will recruit a total of 340 patients with an eating disorder in the university hospital of Montpellier.

* Participation consists of a one-day visit with a multidisciplinary assessment. No action is specific to research. This is the usual management of patients with eating disorders addressed to our department.
* An ancillary study will be proposed, if the patient is addressed by his general practitioner for an annual evaluation. This second visit will be exactly the same as the initial visit.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an eating disorder according to Diagnostic and Statistical Manuel of Mental disorders-V (DSM-V) criteria
* Patient aged from 15 to 65 years
* Patient who performs the day-hospital evaluation
* Patient affiliated to a French social security system
* Patient able to understand the nature, the aim and the methodology of the study
* For minor one of the legal guardians gave his consent

Exclusion Criteria:

* Patient in an unstable somatic state (eg severe metabolic disorder making impossible or unreliable neuropsychological assessments)
* Patient's refusal to participate
* Patient on protective measures (guardianship or trusteeship)
* Pregnant or nursing women. A dosage of beta human chorionic gonadotropin (βHCG) will be performed to ensure the absence of pregnancy.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2017-05-03 (Actual); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Level of functional impairment assessed by the Work and Social Adjustment Scale (WSAS) | Baseline
  We aim to investigate the link between decision-making and daily functioning of patients with eating disorder.

SECONDARY OUTCOMES:
Quality of life assessed by the Eating disorder quality of life (EDQOL) scale. | Baseline
  We aim to investigate the link between quality of life and alteration of cognitive flexibility of patients with eating disorder.
Level of functional impairment assessed by the clinician with the Functional Assessment Staging Test (FAST) scale | Baseline
  We aim to investigate the link between global functioning and alteration of cognitive flexibility of patients with eating disorder.
Quality of life assessed by the Eating disorder quality of life (EDQOL) scale. | Baseline
  We aim to investigate the link between quality of life and alteration central coherence of patients with eating disorder.
Level of functional impairment assessed by the clinician with the FAST scale | Baseline
  We aim to investigate the link between global functioning and alteration central coherence of patients with eating disorder.
Score to decision making test (Iowa gambling task) | At 12 months if patient is included in the ancillary study
  We aim to investigate the prognostic value of decision making abnormalities on the rates of recovery
Score to decision making test (Iowa gambling task) | At 12 months if patient is included in the ancillary study
  We aim to investigate the prognostic value of decision making abnormalities on weight recovery (for anorexic patients)
Score to decision making test (Iowa gambling task) | At 12 months if patient is included in the ancillary study
  We aim to investigate the prognostic value of decision making abnormalities on daily functioning
Score to decision making test (Iowa gambling task) | At 12 months if patient is included in the ancillary study
  We aim to investigate the prognostic value of decision making abnormalities on switch to another subtype of eating disorder
Score to decision making test (Iowa gambling task) | At 12 months if patient is included in the ancillary study
  We aim to investigate the impact of weight recovery on decision making abilities

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Lapeyronie, Montpellier, France

IPD SHARING:
Plan to Share IPD: No